CLINICAL TRIAL: NCT04333095
Title: Regional Blockade of the Sternum With Liposomal Bupivacaine Prior to Incision Decreases Opioid Use in Patients Undergoing Cardiac Surgery (Sternal Block)
Brief Title: Sternal Block With Liposomal Bupivacaine vs. Saline Prior to Incision in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 019-296
Record Dates: First submitted 2020-03-27; First posted 2020-04-03 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Surgery; Pain, Postoperative; Block
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon, coordinator and anesthesiologist on the case are blinded to the block drug. A 2nd (unblinded) anesthesiologist performs the block on the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine Block (Active Comparator): Liposomal Bupivacaine (1.3%) solution (20 mL dose). This solution has demonstrated increased efficacy in prolonged analgesia following injection. This solution will be injected as an ultrasound-guided subpectoral interfacial plane block.
  Interventions: Drug: Liposomal bupivacaine
- Saline Block (Placebo Comparator): Normal saline (0.9%) will be used as the control solution for patients not receiving the liposomal bupivacaine solution. Injection procedure of this solution will be identical to that of the liposomal bupivacaine solution.
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution_#1

INTERVENTIONS:
Drug: Liposomal bupivacaine — Sternal Block during Coronary Artery Bypass Graft Surgery and/or surgical aortic valve replacement through mini- or full sternotomy
  Arms: Liposomal Bupivacaine Block
Drug: Normal Saline Flush, 0.9% Injectable Solution_#1 — Sternal Block during Coronary Artery Bypass Graft Surgery and/or surgical aortic valve replacement through mini- or full sternotomy
  Arms: Saline Block

SUMMARY:
The purpose of this study is to find out what effects (good and bad) that the study medicine called "liposomal bupivacaine" has on subjects that are undergoing a sternotomy. Liposomal bupivacaine solution, is a drug that the doctor will inject before they make the cut through patient's breastbone (sternotomy). Normally pain medicine like this is given right before the surgeon closes up the patient's breastbone, at the end of the surgery. For this study, they want to see if giving the medicine before they make the cut into the patient's breastbone helps their pain. They also want to find out if patients feel less pain after surgery with the study drug than they do with saline and possibly decrease the need for pain medicine. Subjects will be in the study for about 72 hours or until they are discharged from the hospital.

DETAILED DESCRIPTION:
Background:

Prolonged and excessive narcotic usage in the postoperative setting has been linked to multiple complications. Use of complimentary pain management techniques such as regional analgesia can reduce postoperative pain and narcotic usage. This can enhance patient recovery and improve quality of life in the immediate postoperative period. Previous research investigating the benefits of local analgesia during cardiac surgery have been limited by the sparse amount of single-center randomized controlled trials, particularly evaluating the use of para-sternal injections.

Of the available studies, the use of local analgesia injections compared to controls has led to improved pain scores and overall decreased perioperative opioid usage. Studies have shown this efficacy using 0.2% ropivacaine, 0.75% ropivacaine, and 0.53% liposomal bupivacaine all compared to control groups receiving normal saline injections in the para-sternal area. These studies all used injections just prior to sternal closure and no significant evidence is available for the use of ultrasound-guided regional block of the sternum prior to surgical incision. Injection of analgesia prior to surgical incision has been shown to decrease postoperative pain compared to injection after surgical closure.

We hypothesize that injection of 1.3% liposomal bupivacaine and 0.5% bupivacaine (20mL dose) as a sternal block prior to surgical incision will lead to decreased pain and opioid usage in the intraoperative and postoperative setting for patients undergoing upper mini- and median sternotomy compared to controls.

Methods:

This is an investigator-initiated prospective randomized study with an 18-month patient accrual period and patient follow-up period dependent on postoperative length of stay following surgery.

Regional Block: Liposomal Bupivacaine (1.3%) solution (20 mL dose) is proposed for use during this study. This solution has demonstrated increased efficacy in prolonged analgesia following injection. This solution will be injected as an ultrasound-guided subpectoral interfacial plane block.

Normal Saline: Normal saline (0.9%) will be used as the control solution for patients not receiving the liposomal bupivacaine solution. Injection procedure of this solution will be identical to that of the liposomal bupivacaine solution.

Procedures: Patients undergoing a surgical procedure through mini- or full sternotomy will be considered for inclusion in this study. There will be no deviation from routine surgical procedures following injection of para-sternal solution prior to surgical incision.

Data elements:

Patient Characteristics:

1. Age
2. Gender
3. BMI
4. Tobacco use
5. Chronic lung disease
6. Diabetes
7. Hypertension (HTN)
8. Hyperlipidemia (HLD)
9. Ethnicity (Hispanic & not Hispanic)
10. Race (Caucasian, African Americans, Asians and others)
11. Chronic Kidney Disease (CKD)
12. Cerebrovascular accident (CVA)
13. Chronic home non-steroidal anti-inflammatory drug (NSAID) use (excluding acetylsalicylic acid (ASA))

Intraoperative Variables:

1. Type of procedure being performed
2. Prior procedures performed

Postoperative Variables:

Time to extubation, time to ambulation, time to oral diet, return of bowel function, postoperative atrial fibrillation incidence, post op nausea incidence, and intensive care unit (ICU) length of stay (LOS) and overall LOS. Maximum incentive spirometer maximum volume at 24, 48 and 72 hours, Confusion assessment method (CAM) at 24, 48 and 72 hours, post op opioid usage up to 72 hours post op. If additional days of post-op opioid usage is documented in the existing medical record, this may be used also.

Pain scores (Scale 0-10) at 1, 2, 4, 8, 12,24,36,48, 60, and 72 hours after ICU arrival for extubated patients and Clinical Care Pain Observation Tool (CPOT)scores (Scale 0-8) for intubated patients

Adverse Events: Allergic reaction, pneumothorax, pericardial tamponade, vascular injury, hematoma, intravascular injection, wound infection, paresthesia, persistent numbness

Protocol Deviations: If certain data elements are not in the existing medical record and were not collected, this is not a protocol deviation. Nevertheless, all effort will be made to collect these data points.

Risks and Benefits

Risks: The risks are the same as the Standard of Care surgery performed outside this study. This is discussed in the ICF. A confidentiality breach is a risk associated with research. However, all data collection protocols follow HIPAA guidance.

Benefits: If participants receive the drug, they could experience less pain than those that don't receive the drug. However, not all participants are likely to benefit from the proposed research. The investigators will benefit from the knowledge gained, as it will provide deepened insight on the main challenges, advantages and disadvantages of the procedure.

Data Analytic Methods

The mean, standard deviation, median, and interquartile ranges of narcotic usage (in morphine equivalent units) will be reported for each group. The difference of narcotic usage between the two groups will be reported as a single value. Additional variables analyzed in this study include the following:

Patient Characteristics:

1. Age
2. Gender
3. BMI
4. Tobacco use
5. Chronic pain medication usage
6. Diabetes
7. HTN
8. HLD
9. Race & Ethnicity
10. CKD
11. CVA

Intraoperative Variables:

1. Type of procedure being performed
2. Prior procedures performed

Postoperative Variables:

1. Time to extubation
2. Time to ambulation
3. Time to oral diet
4. Postoperative nausea
5. ICU LOS
6. Total LOS
7. Return of bowel function
8. Postoperative atrial fibrillation
9. Maximum spirometry at 24, 48, 72 hours post op
10. CAM at 24, 48, 72 hours post op
11. Pain Scores (Scale 0-10) at 1, 2, 4, 8, 12,24,36,48, 60, and 72 hours after ICU arrival for extubated patients and CPOT scores (Scale 0-8) for intubated patients
12. Post op opioid usage up to 72 hours post op

Standard descriptive statistics will be used throughout (mean, range, standard deviation, and median, IQR), with comparative statistics for normally and non-normally distributed data with p<0.05 considered as significant. For categorical variables, 2 Sample t-test or chi-squared test will be used to determine statistical significance. For continuous variables, logistic regression will be used to determine the value of significance to variables with postoperative outcomes. Depending on the enrollment rate, the stratification of data based on the type of sternotomy (full or mini) could be performed and analyzed respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18 years
2. Undergoing a surgical procedure through mini- or full sternotomy.

Exclusion Criteria:

1. Clinical instability
2. Allergic to liposomal bupivacaine solution or any of its ingredients
3. Maximum-allowed dosage of local analgesia will be exceeded by the injection amount of liposomal bupivacaine used in this study (<50 kg).
4. BMI >45
5. Pregnant or nursing
6. Chronic home opioid usage
7. Left Ventricular Ejection Fraction (LVEF) < 30%
8. Low cardiac output requiring mechanical or inotropic support
9. End-stage renal disease
10. Cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Heart Hospital - Plano, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No
At this point, we do not plan to shared IPD but will share cumulative results in an abstract and manuscript.

REFERENCES:
- [Background] Bignami E, Castella A, Pota V, Saglietti F, Scognamiglio A, Trumello C, Pace MC, Allegri M. Perioperative pain management in cardiac surgery: a systematic review. Minerva Anestesiol. 2018 Apr;84(4):488-503. doi: 10.23736/S0375-9393.17.12142-5. Epub 2017 Oct 12. PMID 29027773
- [Background] Dowling R, Thielmeier K, Ghaly A, Barber D, Boice T, Dine A. Improved pain control after cardiac surgery: results of a randomized, double-blind, clinical trial. J Thorac Cardiovasc Surg. 2003 Nov;126(5):1271-8. doi: 10.1016/s0022-5223(03)00585-3. PMID 14665996
- [Background] Barr AM, Tutungi E, Almeida AA. Parasternal intercostal block with ropivacaine for pain management after cardiac surgery: a double-blind, randomized, controlled trial. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):547-53. doi: 10.1053/j.jvca.2006.09.003. Epub 2006 Dec 22. PMID 17678782
- [Background] Lee CY, Robinson DA, Johnson CA Jr, Zhang Y, Wong J, Joshi DJ, Wu TT, Knight PA. A Randomized Controlled Trial of Liposomal Bupivacaine Parasternal Intercostal Block for Sternotomy. Ann Thorac Surg. 2019 Jan;107(1):128-134. doi: 10.1016/j.athoracsur.2018.06.081. Epub 2018 Aug 28. PMID 30170012
- [Background] Labrum JT 4th, Ilyas AM. Preemptive Analgesia in Thumb Basal Joint Arthroplasty: Immediate Postoperative Pain with Preincision versus Postincision Local Anesthesia. J Hand Microsurg. 2017 Aug;9(2):80-83. doi: 10.1055/s-0037-1603734. Epub 2017 Jun 5. PMID 28867907

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine Block: Liposomal Bupivacaine (1.3%) solution (20 mL dose). This solution has demonstrated increased efficacy in prolonged analgesia following injection. This solution will be injected as an ultrasound-guided subpectoral interfacial plane block.
  Liposomal bupivacaine: Sternal Block during Coronary Artery Bypass Graft Surgery and/or surgical aortic valve replacement through mini- or full sternotomy. We couldn't enroll sufficient mini sternotomies to infer anything statistically so our analysis concentrated on full sterntomies.
- Saline Block: Normal saline (0.9%) will be used as the control solution for patients not receiving the liposomal bupivacaine solution. Injection procedure of this solution will be identical to that of the liposomal bupivacaine solution.
  Normal Saline Flush, 0.9% Injectable Solution_#1: Sternal Block during Coronary Artery Bypass Graft Surgery and/or surgical aortic valve replacement through mini- or full sternotomy. We couldn't enroll sufficient mini sternotomies to infer anything statistically so our analysis concentrated on full sterntomies.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Block | Saline Block
Started | 36 | 34
Full Sternotomy | 32 | 29
Completed (full sternotomy only) | 27 | 25
Not Completed | 9 | 9
Not completed — Protocol Violation | 4 | 0
Not completed — Unblinded anesthesiologist unavailable to give block at the time of surgery | 1 | 4
Not completed — Mini Sternotomy | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine Block | Saline Block | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [65.5 to 74] | 70 [65 to 74] | 70 [65 to 74.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 21 | 17 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 27 | 23 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 1 | 2
  Race: Black | 1 | 1 | 2
  Race: White | 25 | 23 | 48
History of Tobacco Use [Count of Participants; unit: Participants]
  Yes | 8 | 9 | 17
  No | 19 | 16 | 35
Chronic lung disease [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 4
  No | 24 | 23 | 47
  Unknown | 0 | 1 | 1
Hypertension [Count of Participants; unit: Participants]
  Yes | 25 | 20 | 45
  No | 2 | 5 | 7
Hyperlipidemia [Count of Participants; unit: Participants]
  Yes | 23 | 19 | 42
  No | 4 | 6 | 10
Chronic kidney disease [Count of Participants; unit: Participants]
  Yes | 3 | 4 | 7
  No | 24 | 21 | 45
History of cerebrovascular disease [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 4
  No | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Total Postoperative Opioid Measured in Milligram Morphine Equivalent (MME) at 72 Hours
Description: The amount of opioid medications used will be recorded during the routine postoperative course.
Time Frame: Up to 72 hours post-op
Measure: Mean (Standard Deviation); unit: Milligram Morphine Equivalent (MME)
Arm/Group | Liposomal Bupivacaine Block | Saline Block
Number analyzed (Participants) | 27 | 25
Milligram Morphine Equivalent (MME) | 29.4 (16.3) | 25.8 (10.4)

2. Primary Outcome: Intraoperative Opioid Usage Measured in Milligram Morphine Equivalent (MME)
Time Frame: During surgery, up to 7 hours
Measure: Mean (Standard Deviation); unit: Milligram Morphine Equivalent (MME)
Arm/Group | Liposomal Bupivacaine Block | Saline Block
Number analyzed (Participants) | 27 | 25
Milligram Morphine Equivalent (MME) | 114.9 (148) | 124.8 (22.5)

ADVERSE EVENTS:
Time Frame: Until discharged from the hospital, up to 12 days.
Arm/Group | Liposomal Bupivacaine Block | Saline Block
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25

LIMITATIONS AND CAVEATS:
A possible limitation is the overestimation of MME usage in the initial power analysis while calculating the sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT04333095/Prot_SAP_002.pdf